CLINICAL TRIAL: NCT00794911
Title: Quality of Life Therapy for Adults With Hepatitis C Virus and Cirrhosis Awaiting Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, James Rodrigue, Professor of Psychology in the Department of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2007P000171; NCT00794937 (obsolete NCT alias)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2011-03

CONDITIONS: Chronic HCV
Keywords: Liver Transplantation; Quality of Life; Chronic HCV; Hepatitis C Virus; Cirrhosis; Liver disease
MeSH Terms: conditions — Hepatitis C; Fibrosis; Liver Diseases | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- QOLT (Experimental): Quality of Life Therapy (QOLT) 8 weekly individual counseling sessions.
  Interventions: Behavioral: Quality of Life Therapy
- ST (Active Comparator): Supportive Therapy (ST) 8 weekly individual counseling sessions
  Interventions: Behavioral: Supportive Therapy
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Quality of Life Therapy — 8 weekly individual counseling sessions
  Arms: QOLT
Behavioral: Supportive Therapy — 8 weekly individual counseling sessions
  Arms: ST

SUMMARY:
The main purpose of this study is to determine whether psychological intervention is effective in improving quality of life, mood, and relationships among adults with hepatitis C virus and cirrhosis awaiting liver transplantation.

DETAILED DESCRIPTION:
Quality of life (QOL) outcomes are important to all stakeholders in liver transplantation. For patients with end-stage liver disease, QOL is significantly compromised and more data about QOL allows them to make an informed risk-benefit analysis in deciding whether to pursue transplantation. The long-term goal of this research program is to better understand how QOL can be enhanced, to identify the mechanisms underlying QOL changes, to identify which patients benefit most from QOL intervention, and to determine whether QOL benefits can extend beyond transplantation. The objective of this research is to determine the effectiveness, feasibility and applicability of Quality of Life Therapy (QOLT) in treating adults with hepatitis C virus and cirrhosis awaiting liver transplantation. In a recent small, single-center clinical trial, we demonstrated that QOLT can improve QOL, psychological functioning, and social intimacy in patients awaiting lung transplantation. We now seek to examine whether this intervention can be effectively adapted and implemented with adults with hepatitis C virus and cirrhosis awaiting liver transplantation. The central hypothesis is that by targeting improvements in specific life domains, QOLT yields significant clinical benefits in QOL, psychological functioning, and the patient-caregiver relationship. This hypothesis is being tested by pursuing three specific aims: 1) Determine the effectiveness of QOLT; 2) Examine the differential effectiveness of QOLT by race (White, African American); and 3) Assess the feasibility of a multisite R01 application. Under the first aim, adults with hepatitis C virus and cirrhosis awaiting liver transplantation are being randomized to receive QOLT, Supportive Therapy (ST), or Standard Care (SC). Primary outcomes are changes in QOL, psychological functioning, and social intimacy at 1 and 12 weeks post-treatment. Under the second aim, the relationship between race and intervention outcomes will be closely examined. Under the third aim, attrition rates, reasons for attrition, therapist adherence to treatment protocols, and participant satisfaction ratings are being gathered to assess the need for protocol changes prior to developing a larger, multisite clinical trial R01 application. This study is innovative because it is among the first to evaluate a theoretically-driven psychological intervention to specifically improve QOL in the context of hepatitis C virus and cirrhosis and liver transplantation. The research is significant because it is expected to advance and expand understanding of how QOL can be improved in patients with hepatitis C virus and cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 21 and 70 years of age
* Diagnosis of chronic HCV
* Wait-listed for liver transplantation
* Signed informed consent
* Primary caregiver identified as spouse or domestic partner
* Resides within 60 minutes of transplant center
* MELD score < 20

Exclusion Criteria:

* Prior recipient of liver transplantation
* Prior recipient of other solid organ transplantation
* Wait-listed for combined liver-kidney transplantation
* Current substance abuse or dependency
* Currently hospitalized
* Sustained (2 or more consecutive months) MELD score less than or equal to 20
* Current recipient of psychological intervention services
* Substantial cognitive impairment (score of 23 or less on the Mini-Mental State Examination)
* Communication difficulties (speech, hearing) so substantial that they would prevent patient from participating actively in one of the interventions (determined by interviewer rating)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Scores on the following measures at 12 weeks post-intervention: Quality of Life Inventory, SF-36, Liver Disease Quality of Life instrument, CDC's Activity Limitations Module HRQoL-14, Hopkins Symptom Checklist-25, POMS, and Miller Social Intimacy Scale. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James R Rodrigue, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States